CLINICAL TRIAL: NCT07150416
Title: A Single-Arm Clinical Study of Nebulized Inhalation of Recombinant Human p53 Adenovirus Injection (Gendicine) for Treatment of Multiple Ground-Glass Lung Nodules
Brief Title: Nebulized Inhalation of Recombinant Human p53 Adenovirus Injection for Treatment of Multiple Ground-Glass Lung Nodules: A Single-Arm Clinical Study
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Shenzhen SiBiono GeneTech Co.,Ltd (Industry)
Responsible Party: Principal Investigator, Jianxing He, Principal Investigator, Department of Thoracic Surgery, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: rAdp53-LN001
Record Dates: First submitted 2025-08-25; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Multiple Pulmonary Ground-Glass Nodules; Lung Neoplasms; Precancerous Conditions
Keywords: p53 gene therapy; nebulized inhalation; Gendicine; Single-Arm Trial
MeSH Terms: conditions — Lung Neoplasms; Precancerous Conditions

STUDY DESIGN:
Intervention Model Description: This is a single-arm, open-label phase II trial. All enrolled participants will receive the same intervention (nebulized Gendicine®)
Masking Description: This is an open-label study. No masking (blinding) was used as all participants receive the same active intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gendicine Nebulization Arm (Experimental): Participants in this single arm of the study will all receive the active intervention, which is Nebulized Inhalation of Recombinant Human p53 Adenovirus Injection (Gendicine®), at a dose of 1×10¹² VP per session. The treatment will be administered once every three days, for a total of four sessions.
  Interventions: Drug: Recombinant Human Ad-p53 Injection

INTERVENTIONS:
Drug: Recombinant Human Ad-p53 Injection — A replication-deficient recombinant human type 5 adenovirus vector encoding the human wild-type p53 tumor suppressor gene. For this study, it will be administered via nebulized inhalation.

SUMMARY:
This study aims to evaluate the safety and efficacy of nebulized inhalation of Recombinant Human Ad-p53 Injection (Gendicine®) for the treatment of multiple ground-glass lung nodules. This is a single-arm, open-label clinical study conducted at The First Affiliated Hospital of Guangzhou Medical University in China. We plan to enroll approximately 38 patients who have been diagnosed with multiple ground-glass nodules. All participants in this study will receive the nebulized Gendicine® treatment. After the treatment, we will monitor changes in the nodules through regular chest CT scans and record any potential treatment-related reactions to determine if this novel therapy is safe and effective. This study has been approved by the hospital's Ethics Committee.

DETAILED DESCRIPTION:
Background: Ground-glass nodules (GGN) are a common manifestation of early-stage lung adenocarcinoma, and their management strategy (active surveillance or surgical intervention) often presents a dilemma for clinicians and patients. Gendicine® (Recombinant Human Ad-p53 Injection) is a gene therapy product approved in China. Previous studies have shown its ability to induce tumor cell apoptosis and enhance the sensitivity to radiotherapy and chemotherapy in various solid tumors. This study aims to investigate this innovative approach of local administration via nebulized inhalation for treating precancerous lesions or early-stage lung cancer.

Methods: This is a single-arm, open-label, phase II clinical trial utilizing the Simon's optimal two-stage design. The first stage plans to enroll 16 patients. If ≥1 objective response (according to RECIST 1.1 criteria) is observed, the study will proceed to the second stage, with a total planned enrollment of 30 evaluable patients (38 subjects will be recruited accounting for a 20% dropout rate). Participants are patients with multiple ground-glass nodules confirmed by imaging, with at least one nodule pathologically confirmed as malignant. The intervention is nebulized inhalation of Gendicine® at a dose of 1×10¹² VP per time, administered once every three days, for a total of four times. The primary endpoint is the Objective Response Rate (ORR), defined as the proportion of patients achieving Complete Response (CR) or Partial Response (PR) at 6 months post-treatment. Secondary endpoints include safety (assessing adverse events according to CTCAE v5.0), changes in tumor markers, and quality of life scores.

Significance: This study is the world's first clinical trial to explore nebulized inhalation of a gene therapy product for the treatment of lung nodules. Positive results would provide a novel, non-invasive treatment strategy for the very early intervention of lung cancer, potentially delaying or preventing nodule malignancy and avoiding surgical trauma.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. CT scan confirms the presence of multiple ground-glass nodules (GGNs), with at least one nodule measuring between 0.5 cm and 3.0 cm in diameter.
3. At least one GGN is confirmed as malignant or precancerous (e.g., atypical adenomatous hyperplasia, adenocarcinoma in situ) by histopathology or cytology.
4. Life expectancy ≥ 12 weeks.
5. Adequate pulmonary function tests (FEV1 ≥ 70% of predicted value).
6. Signed informed consent.

Exclusion Criteria:

1. Pregnant or lactating women.
2. History of other active malignancies within the past 5 years.
3. Severe cardiac, hepatic, or renal dysfunction (e.g., NYHA class III/IV heart failure, ALT/AST > 3×ULN, Cr > 1.5×ULN).
4. Uncontrolled systemic infection or immunodeficiency diseases.
5. Participation in another interventional clinical trial within 4 weeks prior to enrollment.
6. Known hypersensitivity to any component of the recombinant human p53 adenovirus injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 6 months after the first dose of intervention
  The proportion of participants achieving a best overall response of Complete Response (CR) or Partial Response (PR) according to RECIST 1.1 criteria, based on chest CT scan assessments. CR is defined as the disappearance of all target lesions. PR is defined as at least a 30% decrease in the sum of diameters of target lesions.

SECONDARY OUTCOMES:
Incidence of Treatment-Related Adverse Events | From first dose of study intervention until 30 days after the last dose
  The number and percentage of participants experiencing any treatment-related adverse event (AE), graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in this article will be shared. This includes data on radiological response (CT imaging), safety (adverse events), and baseline characteristics. The data will become available following the publication of the primary results manuscript, with no specified end date. Data will be accessible through a public data repository such as Figshare or ClinicalTrials.gov. Requestors will be required to sign a data access agreement and provide a methodologically sound research proposal for approval by the study steering committee.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and supporting documents will become available after the publication of the primary findings manuscript (anticipated in [年份, e.g., 2026]). Data will be accessible for a minimum of 5 years with no specified end date.
Access Criteria: Data will be available to researchers who provide a methodologically sound proposal. Requestors must sign a data access agreement. Proposals should be directed to the corresponding author or the data access committee at gyfyky_ec@163.com for approval.

REFERENCES:
- [Background] Mazzone PJ, Lam L. Evaluating the Patient With a Pulmonary Nodule: A Review. JAMA. 2022 Jan 18;327(3):264-273. doi: 10.1001/jama.2021.24287. PMID 35040882
- [Background] Aoki T, Hanamiya M, Uramoto H, Hisaoka M, Yamashita Y, Korogi Y. Adenocarcinomas with predominant ground-glass opacity: correlation of morphology and molecular biomarkers. Radiology. 2012 Aug;264(2):590-6. doi: 10.1148/radiol.12111337. Epub 2012 May 31. PMID 22653188
- [Background] Cheng B, Li C, Li J, Gong L, Liang P, Chen Y, Zhan S, Xiong S, Zhong R, Liang H, Feng Y, Wang R, Wang H, Zheng H, Liu J, Zhou C, Shao W, Qiu Y, Sun J, Xie Z, Liang Z, Yang C, Cai X, Su C, Wang W, He J, Liang W. The activity and immune dynamics of PD-1 inhibition on high-risk pulmonary ground glass opacity lesions: insights from a single-arm, phase II trial. Signal Transduct Target Ther. 2024 Apr 19;9(1):93. doi: 10.1038/s41392-024-01799-z. PMID 38637495
- [Background] Pan JJ, Zhang SW, Chen CB, Xiao SW, Sun Y, Liu CQ, Su X, Li DM, Xu G, Xu B, Lu YY. Effect of recombinant adenovirus-p53 combined with radiotherapy on long-term prognosis of advanced nasopharyngeal carcinoma. J Clin Oncol. 2009 Feb 10;27(5):799-804. doi: 10.1200/JCO.2008.18.9670. Epub 2008 Dec 22. PMID 19103729
- [Background] Kastan MB, Canman CE, Leonard CJ. P53, cell cycle control and apoptosis: implications for cancer. Cancer Metastasis Rev. 1995 Mar;14(1):3-15. doi: 10.1007/BF00690207. PMID 7606818
- [Background] Khoo KH, Verma CS, Lane DP. Drugging the p53 pathway: understanding the route to clinical efficacy. Nat Rev Drug Discov. 2014 Mar;13(3):217-36. doi: 10.1038/nrd4236. PMID 24577402
- [Background] Hassin O, Oren M. Drugging p53 in cancer: one protein, many targets. Nat Rev Drug Discov. 2023 Feb;22(2):127-144. doi: 10.1038/s41573-022-00571-8. Epub 2022 Oct 10. PMID 36216888
- [Background] Kruiswijk F, Labuschagne CF, Vousden KH. p53 in survival, death and metabolic health: a lifeguard with a licence to kill. Nat Rev Mol Cell Biol. 2015 Jul;16(7):393-405. doi: 10.1038/nrm4007. PMID 26122615
- [Background] Kim MP, Lozano G. Mutant p53 partners in crime. Cell Death Differ. 2018 Jan;25(1):161-168. doi: 10.1038/cdd.2017.185. Epub 2017 Nov 3. PMID 29099488
- [Background] Mantovani F, Collavin L, Del Sal G. Mutant p53 as a guardian of the cancer cell. Cell Death Differ. 2019 Jan;26(2):199-212. doi: 10.1038/s41418-018-0246-9. Epub 2018 Dec 11. PMID 30538286